CLINICAL TRIAL: NCT02457182
Title: Mindfulness-Based Therapy for Interstitial Cystitis/Bladder Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Gregory Kanter, Urogynecology Fellow, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-141
Record Dates: First submitted 2015-01-08; First posted 2015-05-29 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-01

CONDITIONS: Interstitial Cystitis; Mindfulness; Complementary Medicine; Painful Bladder Syndrome
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-based Stress Reduction (Experimental): Mindfulness-based Stress Reduction (MBSR)
  Interventions: Other: Mindfulness-based Stress Reduction (MBSR); Other: Usual medical therapy
- Usual Care (Placebo Comparator): Usual medical therapy
  Interventions: Other: Usual medical therapy

INTERVENTIONS:
Other: Mindfulness-based Stress Reduction (MBSR)
  Arms: Mindfulness-based Stress Reduction
Other: Usual medical therapy

SUMMARY:
Interstitial cystitis/bladder pain syndrome (IC/BPS) is a poorly understood disease with unreliable treatments. Although it is not known what causes it for certain, we do know that life stressors may make the disease worse or cause flares. Mindfulness Based Stress Reduction (MBSR) is an 8 week class focused on meditation and other techniques that the investigators think may be helpful to people with IC/BPS. This trial will assign participants to an MBSR class or usual care for their IC/BPS to see if the MBSR class would be helpful for their disease.

DETAILED DESCRIPTION:
BACKGROUND/SCIENTIFIC RATIONALE Interstitial cystitis/bladder pain syndrome (IC/BPS) is associated with significant morbidity and poorly understood underlying pathophysiology. IC/BPS comprises a symptom complex defined by the American Urological Association (AUA) as "An unpleasant sensation (pain, pressure, discomfort) perceived to be related to the urinary bladder, associated with lower urinary tract symptoms of more than six weeks duration, in the absence of infection or other identifiable causes"(1). Up to 11% of women are affected by IC/BPS (2), and the disorder may be significantly underdiagnosed (3). A 2008 study (4) indicated that 43% of patients with IC/BPS require multimodal therapy with an average of 7-12 yearly clinic visits at a cost of $9,000/patient. Twenty percent of women report wage losses of >$4000 per year (5). Current theories for the cause of IC/BPS include infectious agents, a defective uroepithelium permeable to toxic substances, structural abnormalities, neurogenic inflammation, increased neurologic sensitivity, or an allergic response involving increased numbers of bladder mast cells (6). Despite these theories, reliable treatments remain elusive. Most IC/BPS treatments target one of these proposed mechanisms, involve trial and error of several therapies (1), and often utilize multiple modalities (7). Treatment success ranges from 47-93% for intravesical instillation to 21-64% for oral therapies, with discontinuation rates up to 80% due to intolerable side effects (1). Efficacious treatments for IC/BPS that apply to a greater proportion of patients with limited side effects are urgently needed.

Mindfulness Based Stress Reduction (MBSR), a Complementary Alternative Medicine (CAM)-based therapy, potentially fulfills this need. The Interstitial Cystitis Association (ICA), a patient-led organization, sponsored a survey of 2100 IC/BPS patients. They reported that 84% had tried CAM therapy and 55% of those surveyed reported that their physicians had recommended CAM (8). According to a 2007 National Health Interview survey (9), CAM is used by 38% of adults in the United States. MBSR has been successfully employed to treat chronic pain syndromes and has been used in disorders such as multiple chemical sensitivity, chronic fatigue syndrome, fibromyalgia (10), and irritable bowel syndrome (IBS) (11). These disorders may coexist in patients with IC/BPS (6). In IC/BPS, increases in stress are positively correlated with increased pain (12); and one study reported that up to 80% of IC/BPS patients found stress reduction decreased their symptoms (8). MBSR was found to be efficacious in the treatment of urgency urinary incontinence, a urinary disorder closely related to IC/BPS (13, 14). While MBSR has shown therapeutic promise in conditions that are similar to or coexist with IC/BPS, and has been rated as helpful by patients suffering from IC/BPS, rigorous randomized clinical trials investigating the efficacy of this intervention are lacking (8).

OBJECTIVES/AIMS/HYPOTHESES Ultimately, the investigators long-term goal is to provide a much-needed treatment for IC/BPS using patient-centered therapy such as MBSR. The objective of this research is to conduct a pilot RCT to explore whether MBSR is acceptable to patients and results in improved symptoms when added to IC/BPS 1st and 2nd-line treatments as recommended in the American Urological Association guidelines (see Table 1). The investigators hypothesize that an 8-week MBSR class will be acceptable to IC/BPS patients and that MBSR used in conjunction with traditional 1st and 2nd line therapies will improve symptoms compared to IC/BPS patients using traditional 1st and 2nd line therapies alone. If this pilot study demonstrates effectiveness and acceptance of MBSR, it would provide data to justify a larger randomized controlled trial. If the investigators' hypothesis is supported with this exploratory study, MBSR, an understudied and potentially underutilized therapy, will expand treatment options for IC/BPS patients. The investigators' aims in pursuit of this goal are; Aim #1: To determine whether the addition of MBSR to 1st and 2nd line therapies as recommended by AUA guidelines improves IC/BPS symptoms as measured by the primary outcome the Global Response Assessment (GRA), as well as the O'Leary-Sant Symptom and Problem Index (OSPI), and Visual Analog (VAS) pain scale. Hypothesis: The investigators hypothesize that MBSR will be an effective treatment for IC/BPS as measured by the validated GRA, O'Leary-Sant and VAS pain scales.

Aim #2: To evaluate whether participation in a structured MBSR class will improve quality of life, sexual function and overall self-efficacy in patients with IC/BPS, based on changes in the Short Form Health Survey (SF-12), Female Sexual Function Index (FSFI), and the Pain Self-Efficacy Scale (SES). Hypothesis: The investigators' hypothesize that MBSR will improve quality of life, sexual function and impressions of self-efficacy as measured by these validated scales

ELIGIBILITY:
Inclusion Criteria:

* Actively utilizing but are incomplete responders to the AUA guideline's 1st or 2nd line therapies
* Non-pregnant women ≥18 years old
* Meets IC/BPS diagnosis by AUA guidelines, OSPI >8
* Negative UA or Urine Culture at time of diagnosis or within 2 months if no change in symptoms over that period
* Able to speak and understand English
* Currently undergoing 1st or 2nd-line treatment as per AUA guidelines, for at least 4 weeks duration

Exclusion Criteria:

* Untreated Urinary tract infection
* Unevaluated Hematuria
* Urinary retention
* Pregnant or lactating women
* History of cystectomy, augmentation cystoplasty or urinary diversion
* History of cystitis potentially due to pelvic radiation or Cytoxan
* Inability to speak and understand English
* Either treatment naïve for IC/BPS or on 3rd line or higher treatment per AUA guidelines

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Kanter, MD, Principal Investigator — Urogynecology Fellow
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597

RESULTS

PARTICIPANT FLOW:
Groups:
- Mindfulness-based Stress Reduction (MBSR): Received usual care continuing current treatments in addition to MBSR
  Mindfulness-based Stress Reduction (MBSR)
  Usual medical therapy
- Usual Care: Received usual care and continue current treatments
  Usual medical therapy
Period: Overall Study
Arm/Group | Mindfulness-based Stress Reduction (MBSR) | Usual Care
Started | 9 | 11
Completed | 8 | 11
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mindfulness-based Stress Reduction (MBSR): Will receive usual care continuing current treatments in addition to MBSR
  Mindfulness-based Stress Reduction (MBSR)
  Usual medical therapy
- Usual Care: Will receive usual care and continue current treatments
  Usual medical therapy
- Total: Total of all reporting groups
Arm/Group | Mindfulness-based Stress Reduction (MBSR) | Usual Care | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (15.2) | 44.4 (13.9) | 45.3 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20
Time with IC diagnosis [Mean (Standard Deviation); unit: years] | 5.0 (5.3) | 3.85 (5.1) | 4.3 (4.96)
Time with IC symptoms [Mean (Standard Deviation); unit: years] | 9.6 (9.9) | 8.9 (7.1) | 9.2 (8.3)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (9.2) | 26.4 (6.0) | 27.1 (7.3)
Race [Number; unit: participants]
  American Indian/Alaskan Native | 0 | 2 | 2
  Asian | 0 | 1 | 1
  Caucasian | 9 | 5 | 14
  Other | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Global Response Assessment (GRA)
Description: The GRA is a 7-point scale, with scores ranging from markedly, moderately or slightly worse to slightly, moderately or markedly improved. This measure is used in many types of research and is not specific to IC/BPS.
Time Frame: Within 2 weeks of 8-week class ending
Measure: Number; unit: participants
Arm/Group | Mindfulness-based Stress Reduction (MBSR) | Usual Care
Number analyzed (Participants) | 8 | 11
participants
  Markedly Improved | 2 | 0
  At least moderately improved | 1 | 3
  At least slightly improved | 7 | 4
  No improvement | 1 | 7

2. Secondary Outcome: O'Leary Sant Symptom Problem Index (OSPI)
Description: The OSPI is a Interstitial cystitis (IC/BPS)-specific scale composed of the symptom index and problem index as well as a total, which sums the symptom and problem scores caused by IC/BPS.
  Symptom scores range from 0-21. Problem scores range from 0-16 Higher scores indicate a worse condition. Total scores range 0-37, with higher scores indicating a worse condition.
Time Frame: Baseline and within 2 weeks of 8-week class ending
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-based Stress Reduction (MBSR) | Usual Care
Number analyzed (Participants) | 8 | 11
units on a scale
  OSPI Total Before | 26.4 (8.1) | 25.4 (6.6)
  OSPI Total After | 18.9 (8.7) | 24.0 (5.6)
  OSPI Symptoms before | 16.1 (5.3) | 15.2 (2.9)
  OSPI symptoms after | 12.5 (4.8) | 14.6 (2.3)
  OSPI Problems before | 10.3 (3.1) | 10.2 (3.9)
  OSPI Problems after | 6.4 (4.0) | 9.4 (3.6)

3. Secondary Outcome: Visual Analog (VAS) Pain Scale
Description: The VAS scale is a 10-point scale ranging from 0 (no pain) to 10 (unbearable pain). 0 is considered better while 10 is considered worse.
Time Frame: Baseline and within 2 weeks of 8-week class ending
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-based Stress Reduction (MBSR) | Usual Care
Number analyzed (Participants) | 8 | 11
units on a scale
  VAS Before | 5.9 (2.4) | 5.7 (2.2)
  VAS After | 4.9 (2.0) | 4.6 (2.1)

4. Secondary Outcome: Short Form Health Survey (SF-12)
Description: The short form health survey (SF-12) is a scale used to evaluate chronic conditions. It is composed of a mental component and physical component. Each is made up of 12 questions totaling a score of 100 points. A zero score indicates the lowest level of health measured and 100 indicates the highest level of health.
Time Frame: Baseline and within 2 weeks of 8-week class ending
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-based Stress Reduction (MBSR) | Usual Care
Number analyzed (Participants) | 8 | 11
units on a scale
  MCS Before | 39.0 (4.5) | 36.6 (6.9)
  MCS After | 47.0 (8.9) | 40.8 (8.1)
  PCS Before | 46.5 (8.6) | 44.1 (9.3)
  PCS After | 46.3 (10.3) | 46.5 (9.3)

5. Secondary Outcome: Female Sexual Function Index (FSFI)
Description: The FSFI measures sexual function. It is composed of 6 individual domain scores (desire, arousal, lubrication, orgasm, satisfaction and pain), which are summed to create a total score. Higher scores indicate better sexual function.
  Ranges:
  Desire 2-10 Arousal 0-20 Lubrication 0-20 Orgasm 0-15 Satisfaction 2-15 Pain 0-15 Total score ranges from 4-95 and is calculated by adding the 6 domains together. Again, higher scores indicate better sexual function.
Time Frame: Baseline and within 2 weeks of 8-week class ending
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-based Stress Reduction (MBSR) | Usual Care
Number analyzed (Participants) | 8 | 11
units on a scale
  Desire before | 2.9 (1.6) | 2.7 (1.4)
  Desire after | 3.5 (1.6) | 2.6 (1.5)
  Arousal before | 2.6 (2.1) | 2.0 (2.2)
  Arousal after | 3.3 (2.3) | 2.3 (2.2)
  Lubrication before | 3.2 (2.7) | 1.6 (2.2)
  Lubrication after | 3.4 (2.4) | 3.1 (2.5)
  Orgasm before | 3.0 (2.7) | 2.2 (2.3)
  Orgasm after | 2.5 (2.5) | 2.3 (2.1)
  Satisfaction before | 2.8 (2.3) | 2.8 (1.9)
  Satisfaction after | 3.8 (1.9) | 3.4 (1.8)
  Pain before | 2.5 (2.4) | 2.1 (2.3)
  Pain after | 3.1 (2.6) | 2.8 (2.4)
  Total before | 16.7 (12.8) | 13.8 (10.9)
  Total after | 19.5 (12.0) | 16.4 (10.9)

6. Secondary Outcome: Pain Self-Efficacy Scale (PSEQ)
Description: The PSEQ is a scale describing how patients rate their abilities to complete daily activities.
  It is a 60 point scale (scores range from 0-60) composed of 10 questions. Higher numbers signify better functioning or less limit by disease. A total score is calculating by summing individual items.
Time Frame: Baseline and within 2 weeks of 8-week class ending
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-based Stress Reduction (MBSR) | Usual Care
Number analyzed (Participants) | 8 | 11
units on a scale
  PSEQ Before | 34.3 (4.5) | 30.8 (10.7)
  PSEQ After | 45.8 (4.9) | 33.5 (9.3)

ADVERSE EVENTS:
Arm/Group | Mindfulness-based Stress Reduction (MBSR) | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No